CLINICAL TRIAL: NCT02560116
Title: The Role of Echocardiographic Contrast (Optison) in Enhancing Tricuspid Regurgitation Spectral Doppler Signals to Assess Pulmonary Artery Systolic Pressures. Correlation With Invasive Measurements Obtained by Right Heart Catheterization
Brief Title: The Role of Echocardiographic Contrast (Optison) in Enhancing Tricuspid Regurgitation Spectral Doppler Signals
Status: Withdrawn | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-283
Record Dates: First submitted 2015-06-24; First posted 2015-09-25 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary artery systolic pressure; Optison
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators aim to correlate noninvasive pulmonary artery systolic pressure (PASP) measurements obtained with and without echocardiographic contrast (Optison) during transthoracic echocardiography (TTE) with those obtained invasively and simultaneously during right heart catheterization, as the gold standard.

DETAILED DESCRIPTION:
In the United States, pulmonary hypertension (PHT) is an increasingly recognized cause of morbidity and mortality.

Echocardiography, due to its widespread use, versatility, portability, noninvasive nature, and safety, is routinely used as the primary method for diagnosis and evaluation of these patients. However, in this very cohort, its accuracy is frequently compromised by poor acoustic windows. The use of echocardiographic contrast (EC) in such patients may increase diagnostic accuracy, eliminate the need for performing more invasive, time-consuming, and expensive tests, and eliminate potential diagnostic and management errors.

Pulmonary Artery Systolic Pressure (PASP) is routinely measured noninvasively with transthoracic echocardiography (TTE) by obtaining the tricuspid regurgitant velocity (TRV) with continuous wave spectral Doppler and applying the modified Bernoulli equation.

The investigators aim to use the FDA approved perflutren-based EC agent Optison to augment inadequate TR CW spectral Doppler envelopes and determine if the TRV and PASP measurements obtained with the use of Optison correlate better with the invasive measurements obtained simultaneously during right heart catheterization as opposed to those measurements obtained without the use of EC.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients (age ≥ 18 years old) undergoing right heart catheterization catheterization laboratory for various clinical indications as part of routine medical care;
* only patients with poor acoustic windows will be included (based on previous studies, body habitus);

Exclusion Criteria:

* atrial fibrillation or other irregular rhythms (bigeminy, frequent ectopy)
* pregnant women
* known allergy to perflutren, blood products, albumin
* patients who cannot receive blood products due to religious beliefs
* evidence of intracardiac right to left shunting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After obtaining informed written consent, investigators will enroll all consecutive patients (age ≥ 18 years old) undergoing right heart catheterization in the catheterization laboratory for various clinical indications as part of routine medical care.
  This will be a prospective and multicenter study. The participating institutions are: North Shore University Hospital (Manhasset, NY), Long Island Jewish Medical Center (New Hyde Park, NY), and Mt Sinai Medical Center (NY, NY).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Noninvasively derived PASP values in patients with versus without Optison enhanced TR continuous wave (CW) spectral Doppler envelopes in patients with technically inadequate studies to PASP measurements obtained invasively and simultaneously | up to 6 months

SECONDARY OUTCOMES:
Continuous wave PASP Doppler Envelope measurements in patients receiving Optison versus conventional non-perflutren based agents (10% air-90% saline mixture). | up to 6 months
  Compare the diagnostic role of Optison versus conventional non-perflutren based agents (10% air-90% saline mixture) in enhancing inadequate TR continuous wave spectral Doppler envelopes. This will be done by measuring the values obtained from echocardiographic and invasive hemodynamics with respect to PASP.
Invasive hemodynamic values in patients who undergo perflutren based EC (Optison) administration on PASP values in patients with normal or elevated PASP. | up to 6 months
Number of patients with adverse events as a measure of safety | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore - LIJ Health System, Manhasset, New York, United States

REFERENCES:
- [Background] Yock PG, Popp RL. Noninvasive estimation of right ventricular systolic pressure by Doppler ultrasound in patients with tricuspid regurgitation. Circulation. 1984 Oct;70(4):657-62. doi: 10.1161/01.cir.70.4.657. PMID 6478568
- [Background] Jeon DS, Luo H, Iwami T, Miyamoto T, Brasch AV, Mirocha J, Naqvi TZ, Siegel RJ. The usefulness of a 10% air-10% blood-80% saline mixture for contrast echocardiography: Doppler measurement of pulmonary artery systolic pressure. J Am Coll Cardiol. 2002 Jan 2;39(1):124-9. doi: 10.1016/s0735-1097(01)01698-9. PMID 11755297
- [Background] Ishii M, Kato H, Inoue O, Takagi J, Akagi T, Miyake T, Sugimura T, Maeno Y, Hashino K, Kawano T. Noninvasive evaluation of systolic pressures of pulmonary artery and right ventricle using contrast-enhanced doppler echocardiography: comparative study using sonicated albumin or glucose solution. Pediatr Cardiol. 1996 May-Jun;17(3):175-80. doi: 10.1007/BF02505208. PMID 8662031
- [Background] Dubourg O, Delorme G, Jondeau G, Chikli F, Clavier H, Valtier B, Terdjman M, Beauchet A, Bourdarias JP. [Simultaneous measurement of systolic pulmonary artery pressure by catheterization and contrast enhancement doppler echocardiography]. Arch Mal Coeur Vaiss. 1993 Dec;86(12):1721-7. French. PMID 8024373
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859